CLINICAL TRIAL: NCT00718172
Title: Viral Kinetics and Liver Gene Expression in Response to Ribavirin and Peginterferon Therapy of Chronic Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080182; 08-DK-0182
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-08-19

CONDITIONS: Hepatitis C, Chronic
Keywords: Ribavirin Pretreatment; Gene Expression; Peginterferon; Hepatitis C; Liver Biopsy; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Adenosine Monophosphate; Ribavirin

INTERVENTIONS:
Procedure: Liver Biopsy
Drug: Peginterferon & Ribavirin for Hepatitis C
Drug: Pre-treatment Ribavirin

SUMMARY:
Up to 120 patients with chronic hepatitis C will be enrolled in a study of viral kinetics and liver gene expression before and during combination therapy with peginterferon and ribavirin. Adult patients with chronic hepatitis C virus (HCV) infection who have compensated liver disease and have not received interferon in the past will be randomized into one of four groups. Groups A and C will undergo liver biopsy before starting peginterferon therapy and Groups B and D will undergo biopsy 6 hours after the initial dose of peginterferon. Furthermore, Groups C and D will receive a run-in period of 4 weeks of ribavirin therapy before starting peginterferon. All patients will receive the standard recommended doses of peginterferon alfa 2a (180 mcg sc weekly) and ribavirin (1000 or 1200 mg daily for genotypes 1, 4-6 and 800 mg daily for genotype 2 and 3) for up to 48 weeks (24 weeks for genotype 2 and 3). All patients in Groups C and D, irrespective of genotype, will be pretreated with ribavirin at a dose of 1000 or 1200 mg, depending on patient body-weight. After the initial peginterferon injection, patients will have blood taken and symptoms recorded at 6, 24, 48, 72 hours and weekly thereafter for four weeks to assess viral kinetic response. Liver biopsy tissue taken before or 6 hours after the initial dose of peginterferon will be assessed by standard light microscopy and also subjected to RNA extraction and microarray analysis of mRNA expression. Patients will be monitored carefully during therapy and tested regularly for HCV RNA levels. Therapy will be given for 48 weeks, but will be discontinued early for patients with genotype 1 infection if HCV RNA levels do not decline by at least 2 log IU/ml by week 12 (lack of an early virological response) or do not decline to undetectable levels by week 24 (lack of HCV RNA clearance). Patients with other genotypes with be treated for a full course of therapy regardless of early responses. After completing therapy, patients will be followed at 4 to 8 week intervals and undergo repeat medical evaluation with liver biopsy 24 weeks after stopping therapy.

The primary clinical criterion for success of therapy is a sustained virological response, as marked by the absence of HCV RNA from serum at least 24 weeks after stopping. The focus of this study, however, will be on viral kinetics comparing patients who were pretreated with ribavirin (Groups C and D) to those who were not (Groups A and B) as well as on gene expression studies assessing the effects of peginterferon on intrahepatic mRNA profiles by comparing Group A and B and the effects of ribavirin by comparing Group A to Group C and Group B to Group D. Results will also be compared between different HCV genotypes. These studies are aimed at assessing the mechanisms of action of peginterferon and ribavirin against HCV and evaluating the basis for the lack of virologic response to combination therapy.

DETAILED DESCRIPTION:
Up to 120 patients with chronic hepatitis C will be enrolled in a study of viral kinetics and liver gene expression before and during combination therapy with peginterferon and ribavirin. Adult patients with chronic hepatitis C virus (HCV) infection who have compensated liver disease and have not received interferon in the past will be randomized into two groups; group A will undergo liver biopsy before starting peginterferon therapy and groups B will undergo biopsy 6 hours after the initial dose of peginterferon. All patients will receive the standard recommended doses of peginterferon alfa 2a (180 mcg sc weekly) and ribavirin (1000 or 1200 mg daily for genotypes 1, 4-6 and 800 mg daily for genotype 2 and 3) for up to 48 weeks (24 weeks for genotype 2 and 3). After the initial peginterferon injection, patients will have blood taken and symptoms recorded at 6, 24, 48, 72 hours and weekly thereafter for four weeks to assess viral kinetic response. Liver biopsy tissue taken before or 6 hours after the initial dose of peginterferon will be assessed by standard light microscopy and also subjected to RNA extraction and microarray analysis of mRNA expression. Patients will be monitored carefully during therapy and tested regularly for HCV RNA levels. Therapy will be given for 48 weeks, but will be discontinued early for patients with genotype 1 infection if HCV RNA levels do not decline by at least 2 log10 IU/ml by week 12 (lack of an early virological response) or do not decline to undetectable levels by week 24 (lack of HCV RNA clearance). Patients with other genotypes with be treated for a full course of therapy regardless of early responses. After completing therapy, patients will be followed at 4 to 8 week intervals and undergo repeat medical evaluation with liver biopsy 24 weeks after stopping therapy.

The primary clinical criterion for success of therapy is a sustained virological response, as marked by the absence of HCV RNA from serum at least 24 weeks after stopping. The focus of this study, however, will be on viral kinetics and gene expression studies assessing the effects of peginterferon on intrahepatic mRNA profiles by comparing Group A and B. Results will also be compared between different HCV genotypes. These studies are aimed at assessing the mechanisms of action of peginterferon and ribavirin against HCV and evaluating the basis for the lack of virologic response to combination therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 years or above, male or female

Presence of HCV RNA (with or without anti-HCV) in serum at levels of at least 10,000 IU/ml.

Willingness to undergo liver biopsy before or 6 hours after an initial injection of peginterferon.

Written informed consent.

EXCLUSION CRITERIA:

Previous adequate treatment with any form of type I interferon (standard alpha interferon, peginterferon, beta interferon). Adequate treatment is considered at least 12 weeks of therapy.

Other antiviral therapy within the last 6 months.

If cirrhosis is present, decompensated liver disease, as marked by bilirubin greater than 4 mg percent, albumin less than 3.0 gm percent, prothrombin time greater than 2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy.

Serum ALT or AST levels greater than 1000 micro/L (greater than 25 times ULN). Such patients will not be enrolled but may be followed until three consecutive determinations are below this level.

Pregnancy or current breastfeeding. In women of child bearing potential or in spouses of such women, inability to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicide, or birth control pills, or an intrauterine device until 6 months after the end of treatment with ribavirin given the potential for teratogenicity.

Significant systemic or major illnesses including congestive heart failure, organ transplantation, serious psychiatric disease or depression, human immunodeficiency virus (HIV) infection, and angina pectoris.

Pre-existing anemia (hematocrit less than 33 percent) or known history of hemolytic anemia. In patients in Groups C and D, liver biopsy will not be performed if hemoglobin levels fall to below 11 g/dl during ribavirin monotherapy. Epopoetin alfa or darbopoietin alfa therapy will be available to achieve an adequate hematocrit if clinically indicated for patients in all groups.

Immunosuppressive therapy with either corticosteroids (more than 5 mg of prednisone daily on a chronic basis) or major immunosuppressive agents (such as azathioprine or 6-mercaptopurine). Patients receiving a short-course of corticosteroids for acute allergic reactions or asthma or chronic obstructive pulmonary disease exacerbations (less than 2 weeks of therapy) will be eligible for the study after 4 weeks off therapy.

Evidence of another form of liver disease in addition to viral hepatitis (for example autoimmune liver disease, Wilson's disease, alcoholic liver disease, hemochromatosis, alpha 1 antitrypsin deficiency). Patients with concomitant non-alcoholic steatohepatitis but no other form of chronic liver disease will not be excluded from this study.

Evidence of coronary artery disease or cerebral vascular disease, including abnormalities on exercise stress testing in patients with defined risk factors who will be screened for evidence of underlying coronary artery disease.

Active substance abuse, such as alcohol, inhaled or injection drugs within the previous year.

Evidence of hepatocellular carcinoma; either alpha-fetoprotein (AFP) levels greater than 200 ng/ml (normal less than 9 ng/ml) and/or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.

Clinical gout.

Active, serious autoimmune disease such as systemic lupus erythematosis, ulcerative colitis, Crohn s disease or rheumatoid arthritis that in the opinion of the investigators might be exacerbated by therapy with alpha interferon.

These exclusion criteria are considered the standard relative contraindications to peginterferon and ribavirin therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-07-11; Study Completion 2014-08-19 (Actual)

PRIMARY OUTCOMES:
Improved viral kinetics with ribavirin pretreatment.

SECONDARY OUTCOMES:
Changes in gene expression during peginterferon and/or ribavirin thereapy, effect of treatment on NK cell function.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rotman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Liang TJ, Rehermann B, Seeff LB, Hoofnagle JH. Pathogenesis, natural history, treatment, and prevention of hepatitis C. Ann Intern Med. 2000 Feb 15;132(4):296-305. doi: 10.7326/0003-4819-132-4-200002150-00008. PMID 10681285
- [Background] Kiyosawa K, Sodeyama T, Tanaka E, Gibo Y, Yoshizawa K, Nakano Y, Furuta S, Akahane Y, Nishioka K, Purcell RH, et al. Interrelationship of blood transfusion, non-A, non-B hepatitis and hepatocellular carcinoma: analysis by detection of antibody to hepatitis C virus. Hepatology. 1990 Oct;12(4 Pt 1):671-5. doi: 10.1002/hep.1840120409. PMID 2170265
- [Background] Hoofnagle JH, Seeff LB. Peginterferon and ribavirin for chronic hepatitis C. N Engl J Med. 2006 Dec 7;355(23):2444-51. doi: 10.1056/NEJMct061675. No abstract available. PMID 17151366
- [Derived] Kim H, de Jesus AA, Brooks SR, Liu Y, Huang Y, VanTries R, Montealegre Sanchez GA, Rotman Y, Gadina M, Goldbach-Mansky R. Development of a Validated Interferon Score Using NanoString Technology. J Interferon Cytokine Res. 2018 Apr;38(4):171-185. doi: 10.1089/jir.2017.0127. PMID 29638206
- [Derived] Serti E, Park H, Keane M, O'Keefe AC, Rivera E, Liang TJ, Ghany M, Rehermann B. Rapid decrease in hepatitis C viremia by direct acting antivirals improves the natural killer cell response to IFNalpha. Gut. 2017 Apr;66(4):724-735. doi: 10.1136/gutjnl-2015-310033. Epub 2016 Jan 4. PMID 26733671
- [Derived] Rotman Y, Noureddin M, Feld JJ, Guedj J, Witthaus M, Han H, Park YJ, Park SH, Heller T, Ghany MG, Doo E, Koh C, Abdalla A, Gara N, Sarkar S, Thomas E, Ahlenstiel G, Edlich B, Titerence R, Hogdal L, Rehermann B, Dahari H, Perelson AS, Hoofnagle JH, Liang TJ. Effect of ribavirin on viral kinetics and liver gene expression in chronic hepatitis C. Gut. 2014 Jan;63(1):161-9. doi: 10.1136/gutjnl-2012-303852. Epub 2013 Feb 8. PMID 23396509